CLINICAL TRIAL: NCT04203628
Title: Evaluation of Four Stool Processing Methods Combined With Xpert MTB/RIF Ultra for Diagnosis of Intrathoracic Paediatric TB
Brief Title: Evaluation of Four Stool Processing Methods Combined With Xpert MTB/RIF Ultra for Diagnosis of Intrathoracic Paediatric TB (TB-Speed - Stool Processing)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: UNITAID (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: C19-34
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Child; Diagnosis; Method; Laboratory
MeSH Terms: conditions — Tuberculosis; Disease

STUDY DESIGN:
Intervention Model Description: Enrolment will have 2 stages. During stage 1 (prospective cohort stage), all consecutive children with presumptive TB enrolled in the TB-Speed HIV or TB-Speed SAM or seen in routine care if ineligible for those two studies will be proposed to participate in the study until we reach the number needed for the evaluation of specificity. All children with presumptive TB will have at least two respiratory samples collected (ES or GA) tested with Ultra and mycobacterial culture. The cohort will be closed once the sample size of presumptive TB children with two negative Ultra results from respiratory samples will be reached.
  During the 2nd phase (enrichment phase), only children with presumptive TB who are Xpert positive on at least one respiratory sample will be proposed to participate in the study in order to complement the number of confirmed TB cases required for the evaluation of the sensitivity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prospective cohort (Experimental): Any child with presumptive TB will be proposed to participate in the study.
  If the child is enrolled in the TB-Speed SAM or HIV studies, the study nurse will collect 2 stool samples then collect information about the clinical examination, chest X-ray, HIV-testing and the mycobacterial culture results as soon as they are available, from the data collected in the TB-speed records since all these procedures are already performed in these studies.
  For children identified from the routine practice, the nurse will collect 2 respiratory samples (sputum or GA) in consecutive children with presumptive TB to be tested using Ultra as done in routine care, record symptoms and refer the child for clinical exam and for chest X-ray. For the purpose of the study, 2 stool samples will be collected to be tested with Ultra. In addition, for study purpose the two respiratory samples will be tested with Mycobacterial culture as this test is not routinely prescribed for TB diagnosis in the study sites
  Interventions: Diagnostic Test: Xpert MTB/Rif Ultra on stool samples; Diagnostic Test: Xpert MTB/Rif Ultra on respiratory sample
- Enrichment cohort (Experimental): Any child with presumptive TB and a positive Xpert result from one respiratory sample (NPA, IS or GA) will be proposed to participate in the study.
  If the child is enrolled in the TB-Speed SAM or HIV studies, the study nurse will collect 2 stool samples then collect information about the clinical examination, chest X-ray, HIV-testing and the mycobacterial culture results as soon as they are available, from the data collected in the TB-speed records since all these procedures are already performed in these studies
  For children identified from the routine care, once enrolled, samples collected as routine practice will be tested with mycobacterial culture in addition to Xpert. If needed an additional respiratory sample will be collected (sputum or GA) and tested with Mycobacterial culture. The nurse will also record symptoms, refer the child for clinical exam and for chest Xray, and collect stool samples. HIV-testing will be offered for children with unknown HIV-status
  Interventions: Diagnostic Test: Xpert MTB/Rif Ultra on stool samples

INTERVENTIONS:
Diagnostic Test: Xpert MTB/Rif Ultra on stool samples — The Xpert MTB/Rif Ultra will be performed on stool samples processed using four different processing methods:
  * Standard sucrose flotation method
  * Optimized sucrose flotation
  * Stool processing kit (SPK)
  * Simple One-step method (SOS)
Diagnostic Test: Xpert MTB/Rif Ultra on respiratory sample — The Xpert MTB/Rif Ultra will be performed on gastric aspirate or expectorated sputum
  Arms: Prospective cohort

SUMMARY:
There is a growing interest for the use of stool samples as an alternative to respiratory samples for the diagnosis of intrathoracic TB in children unable to produce sputum. Unlike respiratory samples, stool samples require processing before molecular testing. Several groups have already evaluated different processing methods. However, it is difficult to know which method has the best accuracy and potential for use at Primary Health Care level, due to the difference in study designs and populations. Therefore, in this study, the investigators propose to evaluate the accuracy of different promising stool processing methods in the same population within the same study with an adapted design. Furthermore, no study has so far evaluated for stool testing the new Xpert MTB/RIF Ultra cartridge that has a lower level of detection than the previous Xpert MTB/RIF cartridge. The investigators propose to evaluate the accuracy of Xpert MTB/RIF Ultra (Ultra) performed on stool samples collected from children with presumptive TB and processed using four different processing methods (Standard sucrose flotation method, optimized sucrose flotation method, SPK, and SOS) against bacteriological results from respiratory specimens and to perform a head-to-head comparison of the diagnostic accuracy and feasibility of these different methods in Uganda and Zambia. The selection of processing methods was based on accuracy results, degree of simplification allowing their introduction at PHC level, and finding from the TB-Speed in-vitro stool processing study. The standard sucrose flotation method is kept to assess if results obtained with the optimised sucrose-flotation method in our in-vitro study can be reproduced in-vivo

DETAILED DESCRIPTION:
This is a diagnostic study evaluating the diagnostic accuracy of the Ultra assay in stools with a two-stage sequential design starting as a cohort of children with presumptive TB enriched in a second stage with Ultra positive TB cases on respiratory sample. It is both an ancillary to the TB-Speed HIV (C18-27) and the TB-Speed SAM (C18-28) studies and a study enrolling children from routine not enrolled in those two studies.

This design was chosen to be able to evaluate the sensitivity and specificity of the Ultra assay in a smaller sample size that is usually required by a "classical" prospective cohort design and avoiding the bias of overestimation of the sensitivity classically associated with the case-control design. In order to quickly generate data on appropriate stool processing method, and to contribute to the planned WHO recommendations for stool Ultra testing (expected 2nd semester 2020), a two-stage sequential design will be used. Indeed, knowing that on average only 10-15% of children with presumptive TB in a community-based setting will be confirmed, in order to reach the sample size of confirmed cases for the evaluation of sensitivity, 7 to 10 times more children with presumptive TB would need to be enrolled in a prospective design. On the other hand, the number of children with presumptive TB not confirmed with TB for the estimation of the specificity would be reached much earlier. In addition, based on the previous study results, it is known that the specificity of Xpert MTB/RIF assay in stool is high (99% CI:98-99), which would result in a relatively small sample size to evaluate the specificity of the Ultra in stools.

During the first stage, the investigators will offer to join all consecutive presumptive TB cases presenting at study sites to estimate specificity with the expected precision and calculate a preliminary sensitivity estimate. During the second stage, the investigators will keep enrolling only those from TB Speed studies and routine care who are Xpert positive on respiratory samples in order to estimate sensitivity with the expected precision.

This two-stage sequential design first estimating specificity then sensitivity has been described by Wruck et al. as an efficient way of validating diagnostic tests when the prevalence of the disease is low. It would not be feasible to consecutively enrol all children with presumptive TB to describe an expected sensitivity of 60% with 10% precision as this would require over 900 patients, of which, approximately 800 would be culture negative. In the two-stage process described by Wruck, only reference standard positive samples from the original population are selected in stage 2. The investigators adapted this design to the TB context as culture results will only be available after enrollment (and if the child is positive, only after the child has started treatment), hence selecting only those who are Ultra positive on respiratory samples for the second cohort as a way of enriching the study population with a subpopulation that has a higher TB prevalence probability, before their true disease status is confirmed. Other comparable diagnostic studies have either used greater resources to include larger samples sizes or have resorted to reporting imprecise estimates of sensitivity. To our knowledge, this is a relatively unique approach to study design for accuracy studies, with few published examples.

With such design, there should be no bias on the evaluation of the specificity similarly to a classical prospective design because this evaluation will be done among consecutively enrolled children with presumptive TB only. The sensitivity estimates may not be generalizable to all culture confirmed TB children due to the sampling approach. Xpert positive children will be more likely to have higher biological loads, causing a possible inflation of the sensitivity. However, the results will provide valuable information on variations of sensitivities of the different stool processing methods within this population.

An interim analysis will be carried out after the completion of the prospective cohort in order to describe specificity and preliminary results of the sensitivity and the agreement between the processing methods. The recruitment of participants will not be put on hold during the interim analysis. A final analysis will be conducted at the end of the study to describe sensitivity as well as the secondary end points.

ELIGIBILITY:
Inclusion Criteria for the prospective cohort:

1. Children < 15 years old
2. Presumptive intra-thoracic TB based on at least one criterion among the following:

   * Persistent cough for more than 2 weeks
   * Persistent fever for more than 2 weeks
   * Recent failure to thrive (documented clear deviation from a previous growth trajectory in the last 3 months or Z score weight/age < 2)
   * Failure of broad-spectrum antibiotics for treatment of pneumonia
   * Suggestive CXR features

   OR History of contact with a TB case and any of the symptoms listed under point 2 with shorter duration (< 2 weeks) if the child is HIV infected or presents with SAM.
3. Signed informed consent by parent or guardian and assent signed by children ≥ 7 years old

Inclusion Criteria for the enrichment cohort:

1. Children < 15 years old
2. Presumptive TB based on at least one criterion among the following:

   * Persistent cough for more than 2 weeks
   * Persistent fever for more than 2 weeks
   * Recent failure to thrive (documented clear deviation from a previous growth trajectory in the last 3 months or Z score weight/age < 2)
   * Failure of broad-spectrum antibiotics for treatment of pneumonia
   * Suggestive CXR features

   OR History of contact with a TB case and any of the symptoms listed under point 2 with shorter duration (< 2 weeks) if the child is HIV infected or presents with SAM.
3. One positive Xpert (MTB/Rif or Ultra) result from at least one respiratory sample: sputum, NPA or GA
4. Signed informed consent by parent or guardian and assent signed by children ≥ 7 years old

Exclusion Criteria for prospective and enrichment cohorts:

1. > 5 days of antituberculosis treatment in the last 3 months
2. History of tuberculosis preventive therapy in the last 3 months
3. Confirmed extrapulmonary TB only

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 215 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
Sensitivity and sensibility of Ultra on stool | 8 weeks
  Sensitivity and specificity of Ultra on stool using TB culture reference standard (LJ and MGIT) in two respiratory samples (two sputums or two gastric aspirates according the age of the child).

SECONDARY OUTCOMES:
Per-protocol analysis of diagnostic accuracy of Ultra on stool using TB culture reference standard | 8 weeks
  Per-protocol analysis of sensitivities and specificities of Ultra on stool using TB culture reference standard (LJ ans MGIT) in respiratory sample, excluding invalid Ultra results and contaminated culture results from analysis.
Head-to-head comparisons | 8 weeks
Sensitivities and specificities of each sampling method | 8 weeks
  * Sensitivities and specificities of each sampling method using TB culture reference standard
  * Sensitivities and specificities of each sampling method using the TB composite reference standard as defined by the Expert Committee (Clinical Case Definition for Classification of Intrathoracic Tuberculosis in Children)
Proportion of Ultra "trace" results in stools out of the number of stools tested with Ultra | 8 weeks
Proportion of Ultra semi-quantitative results "very low"; "low"; "medium" and "high" in stool | 8 weeks
Proportion of invalid Ultra results from stool out of the number of stools tested with Ultra | 8 weeks
Proportion of Rifampicin resistant results on Ultra (stool and respiratory), LPA and DST | 8 weeks
Stratification of characteristics and laboratory results by age groups (≤2 years and > 2 years) | 8 weeks
Proportion of children successfully providing a stool sample | 8 weeks
Relative gain of the 2nd stool sample as compared to the 1st one | 8 weeks
  Relative gain of the 2nd stool sample as compared to the 1st one as measured by the number of additional positive results obtained from the addition of the 2nd sample as compared to the results of the first sample only
Feasibility assessment of the stool processing methods | 25 months
  Feasibility assessment by laboratory technician of their perception of ease of use, safety and suitability to low primary health care setting using a questionnaire and a standard "Ease of use score".
  The assessment will be divided into 2 parts:
  * General characteristics of the stool processing method will be scored according to a rating system laying on 10 criteria describing the ease of use. The score range from 1 to 50, each criteria being scored from 1 to 5. A low score reflects the lowest levels of complexity of sample processing procedures.
  * Characteristic related to the opinion of the laboratory technician (rapidity and ease of performance, quality of instruction sheet, perceived feasibility at each step). The opinion of all study laboratory technicians will be assessed independently and using a short self-administered questionnaire containing open and multiple-choice questions

CONTACTS AND LOCATIONS:
Overall Officials: Maryline Bonnet, MD, PhD, Principal Investigator — Institut de Recherche pour le Développement (IRD) Montpellier, France; Olivier Marcy, MD, PhD, Principal Investigator — University of Bordeaux, France; Eric Wobudeya, MD, PhD, Principal Investigator — MU-JHU Care Ltd, Kampala, Uganda
Locations (3):
- Mbarara Regional Hospital, Mbarara, Uganda
- Zambia (2):
  - Lusaka University Teaching Hospital, Lusaka
  - Arthur Davidson Children Hospital, Ndola

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available after de-identification
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Access to data will be given after the publication of the main study results based on global data.
Access Criteria: Data can be requested by members or partners of the TB-Speed consortium or by external research groups.
  They can be used for secondary analyses of the TB-Speed project, country specific analyses, contribution to individual data meta-analysis and analyses that are not related to the research thematic of TB-Speed project.
  The request for access to data will need to be sent to the Publication Committee accompanied by a concept paper describing the objectives of the analysis/study, how the data will be used, the list of data or material requested and how the original contributors will be credited.
  Once the application is approved, data will be released under a data and/or material sharing agreement that secures the term of use.

REFERENCES:
- [Derived] Lounnas M, Masama EN, Beneteau S, Kasakwa K, Kaitano R, Nabeta P, Ruhwald M, De Haas P, Tiemersma EW, Nduna B, Nicol MP, Eyangoh S, Wobudeya E, Mwanga-Amumpaire J, Chabala C, Marcy O, Bonnet M; TB-Speed Stool Study Group. Centrifuge-free stool processing methods for Xpert MTB/RIF Ultra tuberculosis diagnosis in children in Uganda and Zambia: an observational, prospective, diagnostic accuracy study. Lancet Microbe. 2025 Aug;6(8):101055. doi: 10.1016/j.lanmic.2024.101055. Epub 2025 Jun 23. PMID 40570871
- See also: TB-Speed project official website — https://www.tb-speed.com/